CLINICAL TRIAL: NCT00851734
Title: A Phase 1 Dose-Escalation Study To Assess the Safety and Tolerability of LX214 Ophthalmic Solution in Healthy Volunteers, Followed By an Open-Label Evaluation of LX214 Ophthalmic Solution in Patients With Keratoconjunctivitis Sicca
Brief Title: A Dose-Escalation Study to Assess the Safety and Tolerability of LX214 Ophthalmic Solution in Healthy Volunteers, Followed by an Open-Label Evaluation of LX214 in Patients With Keratoconjunctivitis Sicca (KCS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lux Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LX214-01
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Keratoconjunctivitis Sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LX214 0.02% (Experimental): LX214 ophthalmic solution 0.02%
  Interventions: Drug: voclosporin ophthalmic solution
- LX214 0.2% (Experimental)
  Interventions: Drug: voclosporin ophthalmic solution
- placebo (Placebo Comparator): placebo
  Interventions: Drug: voclosporin ophthalmic solution

INTERVENTIONS:
Drug: voclosporin ophthalmic solution — 0.02%, 0.2% t.i.d. or b.i.d.

SUMMARY:
This is a first-in-man study for the purpose of determining the safety and tolerability of LX214 ophthalmic solution in healthy volunteers and in patients with dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease as determined by a physical examination, clinical laboratory evaluation, and an ECG
* Schirmer's I Test ≥ 10mm/5 minutes with anesthesia
* Corrected Snellen acuity of 20/40 or better in both eyes

Exclusion Criteria:

* Subjects diagnosed with any ocular disease other than refraction error
* Subjects with intraocular pressure >21 mmHg
* Use of a contact lens within 7 days prior to administration of the first dose
* Subjects with history of ocular surgery
* Subjects with a history of laser refractive surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
ocular irritation | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Product Investigations, Conshohocken, Pennsylvania, United States